CLINICAL TRIAL: NCT03183791
Title: RELAXaHEAD for Headache Patients (Phase I)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 17-00525
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2020-02

CONDITIONS: Headache; Migraine; Multiple Sclerosis
MeSH Terms: conditions — Headache; Migraine Disorders; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RELAX group (Experimental)
  Interventions: Behavioral: RELAXaHEAD app
- Monitored Usual Care (MUC) group (Active Comparator)
  Interventions: Behavioral: Monitored Usual Care (MUC)

INTERVENTIONS:
Behavioral: RELAXaHEAD app — The Research Volunteers (RV) will explain the rationale for PMR and load the RELAXaHEAD app onto the patients' smartphones. The RV will review the app with the subject, focusing on user knowledge, usability, and engagement. The patient will perform a 15 minute session of PMR during the study enrollment and discuss the optimal time and place to practice PMR at home. Subjects will also be taught to enter their headache log daily on the app.
  Arms: RELAX group
Behavioral: Monitored Usual Care (MUC) — The Research Volunteers (RV) will load the app onto the patients' smartphones but the PMR component will be blocked on the version of the app that the MUC patients receive.
  Subjects will be taught to enter their headache log daily on the app.
  Arms: Monitored Usual Care (MUC) group

SUMMARY:
The goal of this research is to assess the utility of smartphone-based progressive muscle relaxation (PMR) for the treatment of headaches. While there are many commercially available electronic diary and mind-body intervention apps for headache, there is little data showing their efficacy. RELAXaHEAD app incorporates the electronic PMR that was successfully used in an earlier epilepsy study and beta tested with headache specialist and migraine patient input. It also is an electric headache diary. This 2-arm randomized controlled study will evaluate the feasibility and acceptability of RELAX for use with headache patients. One arm will be the RELAX group (the RELAXaHEAD app) and the other arm will be a monitored usual care (MUC) group (this group receives standard of care and uses the electronic daily symptom reporting diary). The goals are to assess the feasibility and adherence of the RELAX intervention in persons with headache (Aim 1) and to gather exploratory data on the effects of the RELAX intervention on headache related outcome measures (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* Meets migraine criteria based on International Classification of Headache Disorders (ICHD) 3 beta (based on questions in RedCap
* 4 or more headache days per month

Exclusion Criteria:

* Patients who have had Cognitive Behavioral Therapy, Biofeedback or other Relaxation Therapy for Migraine in the past year
* Cognitive deficit or other physical problem with the potential to interfere with behavioral therapy
* Alcohol or other substance abuse as determined by self-report or prior documentation in the medical record
* Opioid or barbiturate use 10+ days a month
* Unable or unwilling to follow a treatment program that relies on written and audio recorded materials
* Not having a smartphone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Number of days spent logging headache data as determined by entries into the RELAXaHEAD app | 90 Days
  Measure of feasibility
Number of days spent doing PMR as determined with the backend analytics in the RELAXaHEAD app backend analytics in the RELAXaHEAD app | 90 Days
  Measure of feasibility
Minutes/day spent doing PMR as determined with the backend analytics in the RELAXaHEAD app | 90 Days
  Measure of feasibility
Satisfaction using Likert scale questions on RELAXaHEAD usability, content, and functionality | Baseline
  Measure of acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Mia Minen, MD, Principal Investigator — New York Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No